CLINICAL TRIAL: NCT07150806
Title: Progressive/Recurrent Intracranial Meningioma Treated With SSTR-Targeted Alpha Emitter RYZ101 (PRIMe-STAR)
Brief Title: RYZ101 for the Treatment of Progressive or Recurrent Intracranial Meningioma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joshua Palmer (Other)
Collaborators: RayzeBio, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Joshua Palmer, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-24368; NCI-2025-06045 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Meningioma
MeSH Terms: conditions — Meningioma | interventions — Specimen Handling; Ga(III)-DOTATOC; gallium Ga 68 dotatate; Arginine; Lysine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (RYZ101) (Experimental): Patients receive RYZ101 IV and amino acids, with L-arginine and L-lysine, IV on day 1 of each cycle. Cycles repeat every 8 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients receive gallium Ga 68-DOTATATE IV and undergo PET scan or SSTR PET scan, CT scan, MRI and undergo blood and urine sample collection and may undergo echocardiography or MUGA scan throughout the study.
  Interventions: Drug: Actinium Ac 225 DOTATATE RYZ101; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Radiation: Gallium Ga 68-DOTATATE; Drug: L-lysine/L-arginine-containing Amino Acid; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Procedure: Somatostatin Receptor Positron Emission Tomography

INTERVENTIONS:
Drug: Actinium Ac 225 DOTATATE RYZ101 — Given IV
  Other Names: 225Ac-DOTA-TATE RYZ101; 225Ac-Oxodotreotide; Actinium Ac 225-Dotatate RYZ101; ACTINIUM AC-225 DOTATATE; RYZ 101; RYZ-101; RYZ101
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Radiation: Gallium Ga 68-DOTATATE — Given IV
  Other Names: (68)Ga-DOTA-TATE; 68Ga-DOTA-0-Tyr3-Octreotate; 68Ga-DOTATATE; Gallium Ga 68 Oxodotreotide; Gallium Oxodotreotide Ga-68; Gallium-68 DOTA-DPhe1, Tyr3-octreotate
Drug: L-lysine/L-arginine-containing Amino Acid — Given IV
  Other Names: Amino Acid Renal Protectant Solution; Amino Acid Solution-containing L-lysine and L-arginine; Intravenous L-lysine/L-arginine-containing Amino Acid Solution; L-lysine/L-arginine AA Solution; Lysine-Arginine Amino Acid Solution; Lysine/Arginine Amino Acid Solution; Radioprotective Amino Acid Solution
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Somatostatin Receptor Positron Emission Tomography — Undergo SSTR PET scan
  Other Names: SSTR-PET

SUMMARY:
This phase I/II tests the safety, side effects, best dose and how well giving RYZ101 works for the treatment of patients with intracranial meningioma that is growing, spreading, or getting worse (progressive) or that has come back after a period of improvement (recurrent). RYZ101 is a radioactive drug. It binds to a protein called somatostatin receptor, which is found on some neuroendocrine tumor cells. Lutetium Lu 177-dotatate builds up in these cells and gives off radiation that may kill them. It is a type of radioconjugate and a type of somatostatin analog. Giving RYZ101 may be safe, tolerable and/or effective in treating patients with progressive or recurrent intracranial meningioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the efficacy of 225Ac-DOTATATE (RYZ101) therapy in the treatment of patients with progressive or recurrent grade 1-3 intracranial meningioma as measured by the progression free survival at 6 months.

SECONDARY OBJECTIVES:

I. To evaluate the objective response rate (ORR) by standard of care brain magnetic resonance imaging (MRI) at 6 months and gallium Ga 68-DOTATATE (68Ga-DOTATATE) positron emission tomography (PET) imaging at 1 year.

II. To determine the overall survival (by grade cohort) in patients with progressive / recurrent meningioma during or after treatment with RYZ101.

III. To determine the progression-free survival (by grade cohort) in patients with progressive / recurrent meningioma during or after treatment with RYZ101.

IV. To determine the toxicity rate in patients with progressive / recurrent meningioma during or after treatment with RYZ101.

V. To perform semiquantitative analysis of PET standardized uptake value (SUV) uptake and compare to the background for treatment response assessment and as a potential biomarker of response and prognosis.

OUTLINE:

Patients receive RYZ101 intravenously (IV) and amino acids, with L-arginine and L-lysine, IV on day 1 of each cycle. Cycles repeat every 8 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients receive Ga 68-DOTATATE IV and undergo PET scan or somatostatin receptor (SSTR) PET scan, computed tomography (CT) scan, MRI and undergo blood and urine sample collection and may undergo echocardiography or multigated acquisition (MUGA) scan throughout the study.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of age > 18 years
* Patients with 68Ga-DOTATATE positive recurrent or progressive meningiomas, any World Health Organization (WHO) grade, who have progressed after first line treatment.

  * For Grade I meningioma, patients must have either:

    * Progressive disease after at least surgical resection and radiotherapy, as defined as an increase in size of the measurable primary lesion (bidirectional area) on imaging by 25% or more between scans separated by no more than 12 months; or
    * Progressive residual tumor after maximal safe resection, located at or near critical organs at-risk and considered to be high-risk for radiation injury by the treating investigator. Prior external beam radiotherapy is not required for these subjects.
  * For Grade II or III meningioma, subjects must have either:

    * Progressive disease after at least surgical resection and radiotherapy, as defined as an increase in size of the measurable primary lesion (bi-directional area) on imaging by 25% or more between scans separated by no more than 12 months or
    * Residual measurable disease after prior surgery without requirement of progression, or
    * Unsuitable for, or decline other standard of care treatment.
* Positive 68Ga-DOTATATE uptake on PET/CT at baseline, defined as target lesion uptake higher than the background with SUV ratios adjusted to the liver uptake (Krenning score ≥ 2)
* Presence of measurable disease defined as at least one lesion measuring ≥ 5 mm in at least one dimension by contrast-enhanced MRI performed within 30 days prior to study registration
* Multifocal disease allowed but limited to ≤ 3 measurable intracranial lesions on the most recent post-contrast MRI
* There is no limit on the number of prior surgeries, radiation therapy, radiosurgery, systemically administered therapeutic agents or theranostic agents
* For patients treated with external beam radiation, interstitial brachytherapy or radiosurgery, an interval ≥ 24 weeks must have elapsed from completion from these therapies to registration unless there is histopathologic confirmation of recurrent tumor or there is new enhancing tumor outside the radiation field (beyond the high dose region or the 80% isodose line)
* An interval of ≥ 28 days (or 5 half-lives, whichever is shorter) from prior cytotoxic chemotherapy (6 weeks from nitrosoureas), biologic agent, investigational agent or any other systemic agent prescribed for the purpose of treating meningioma
* An interval of ≥ 28 days from craniotomy and ≥ 7 days from stereotactic biopsy
* Patients must be willing and able to undergo regular MRI scans of the brain
* Patients must have recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade ≤ 1 or pretreatment baseline from clinically significant adverse events related to prior therapy (exclusions include alopecia, laboratory values listed per inclusion criteria, lymphopenia, sensory neuropathy ≤ grade 2, or other ≤ grade 2 not constituting a safety risk based on the investigator's judgment)
* Any neurological symptoms must be stable for at least 28 days prior to enrollment and patients should not require escalating doses of steroids to control neurological symptoms (stable low dose maintenance steroids at ≤ 8 mg dexamethasone or equivalent are allowed)
* Sufficient renal function, as evidenced by creatinine clearance (CrCl) ≥ 60 mL/min calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
* Hemoglobin concentration ≥ 5.0 mmol/L (≥ 8.0 g/dL)

  * Note: Colony-stimulating factors, platelet-production stimulators and/or transfusions within 4 weeks prior to screening and first dose of study treatment are not permitted to meet these criteria
* Absolute neutrophil count (ANC) ≥ 1000 cells/µL (≥ 1000 cells/mm^3)

  * Note: Colony-stimulating factors, platelet-production stimulators and/or transfusions within 4 weeks prior to screening and first dose of study treatment are not permitted to meet these criteria.
* Platelets > 100 × 10^9/L (100 × 10^3/mm^3)

  * Note: Colony-stimulating factors, platelet-production stimulators and/or transfusions within 4 weeks prior to screening and first dose of study treatment are not permitted to meet these criteria.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN) (or ≤ 5 × ULN if presence of liver metastases)
* Total bilirubin ≤ 3 × ULN
* Serum albumin ≥ 3.0 g/dL
* Adequate coagulation function, defined by international normalized ratio (INR) or prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN, unless subject is receiving anticoagulant therapy and PT or aPTT is within therapeutic range of intended use of anticoagulants
* For women of childbearing potential (WOCBP):

  * Negative pregnancy test within 48 hours prior to the first dose of study treatment
  * Agreement to use barrier contraception and a second form of highly effective contraception while receiving study treatment and for 7 months following their last dose of study treatment. Alternatively, total abstinence is also considered a highly effective contraception method when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

A woman is considered to be of childbearing potential if she is postmenarche, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea [no menstrual bleeding of any kind, including menstrual period, irregular bleeding, spotting, etc.] with no identified cause other than menopause), and has not undergone surgical sterilization (total hysterectomy, or bilateral tubal ligation or bilateral oophorectomy at least 6 weeks before first dose of study treatment)

* Sexually active male subjects must use a condom during intercourse while receiving RYZ101 and for at least 120 days after the last dose of the study treatment and should not father a child during this period.

  * Male study subjects whose sexual partners are WOCBP must also agree to use a second form of highly effective contraception while receiving RYZ101 and for at least 4 months following their last dose. Alternatively, total abstinence is also considered a highly effective contraception method when this is in line with the preferred and usual lifestyle of the subject.
  * Vasectomized men are also required to use a condom during intercourse, including with a male partner, to prevent delivery of the drug via seminal fluid.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* Received radiation therapy to the brain in last 24 weeks
* History of hypersensitivity or allergy to Actinium Ac-225 (225Ac), Gallium Ga 68 (68Ga), Copper Cu 64 (64Cu), octreotate, or any of the excipients of DOTATATE imaging agents
* Prior radiopharmaceutical therapies (RPT), including radioembolization
* Prior solid organ or bone marrow transplantation
* Any toxicities from prior treatments that have not recovered to CTCAE grade ≤1, except for alopecia
* Significant cardiovascular disease, defined as:

  * New York Heart Association (NYHA) Class ≥ II heart failure.
  * Known left ventricular ejection fraction (LVEF) < 50%.
  * History of myocardial infarction, acute coronary syndrome, or coronary angioplasty/stenting/bypass within the last 6 months.
  * QT interval corrected for heart rate using Fridericia's formula (QTcF) > 470 ms, demonstrated by the average value of 3 consecutive electrocardiograms (ECGs).
  * Resistant hypertension, defined as persistent uncontrolled blood pressure (BP) > 140/90 mmHg while on optimal doses of at least 3 antihypertensive medications with 1 being a diuretic. Patients with baseline hypertension may be eligible after initiation of antihypertensive therapy
* Uncontrolled diabetes mellitus as defined by hemoglobin A1C (HgB A1c) > 8% in patients with known diagnosis of diabetes mellitus)
* Liver cirrhosis
* Pregnancy or lactation
* Unable to understand or unwilling to sign an Institutional review board approved written informed consent document
* Current somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | At 6 months
  Defined as survival without progression of disease (progressive disease, based on Response Assessment in Neuro-Oncology Criteria [RANO] 2.0 criteria) or death. Kaplan-Meier analyses will be used to estimate PFS.

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 6 months and 1 year
  Assessed by standard of care brain magnetic resonance imaging (MRI) at 6 months and gallium Ga 68-DOTATATE positron emission tomography (PET) at 1 year. ORR defined as the best response including complete response, partial response or stable disease per RANO 2.0 criteria.
Overall survival (OS) | From the date of trial enrolment to date of death, up to 2 years
  Kaplan-Meier analyses will be used to estimate OS.
Incidence of adverse events | Up to 2 years
  The number and type of adverse events will be summarized, using the NCI's Common Toxicity Criteria for Adverse Events, version 5.0 (CTCAE V.5.0).
PET standardized uptake value uptake | Up to 2 years
  To compare to the background for treatment response assessment and as a potential biomarker of response and prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Palmer, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu